CLINICAL TRIAL: NCT03608631
Title: Phase I Study of Mesenchymal Stromal Cells-Derived Exosomes With KrasG12D siRNA for Metastatic Pancreas Cancer Patients Harboring KrasG12D Mutation
Brief Title: iExosomes in Treating Participants With Metastatic Pancreas Cancer With KrasG12D Mutation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0126; NCI-2018-01441 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0126 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-07-16; First posted 2018-08-01 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: KRAS NP_004976.2:p.G12D; Metastatic Pancreatic Adenocarcinoma; Pancreatic Ductal Adenocarcinoma; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (iExosomes) (Experimental): Participants receive mesenchymal stromal cells-derived exosomes with KrasG12D siRNA IV over 15-20 minutes on days 1, 4, and 10. Treatment repeats every 14 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Participants who respond may continue 3 additional courses.
  Interventions: Drug: Mesenchymal Stromal Cells-derived Exosomes with KRAS G12D siRNA

INTERVENTIONS:
Drug: Mesenchymal Stromal Cells-derived Exosomes with KRAS G12D siRNA — Given IV
  Other Names: MSC-derived Exosomes with KrasG12D siRNA (SY); KrasG12D siRNA-loaded Mesenchymal Stromal Cells-derived Exosomes (SY)

SUMMARY:
This phase I trial studies the best dose and side effects of mesenchymal stromal cells-derived exosomes with KrasG12D siRNA (iExosomes) in treating participants with pancreatic cancer with KrasG12D mutation that has spread to other places in the body. iExosomes may work better at treating pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the maximum tolerated dose (MTD) of mesenchymal stem cell (MSC)-derived exosomes loaded with small interference RNA (siRNA) against KrasG12D (iExosomes) in metastatic pancreatic ductal adenocarcinoma (PDAC) patients with KrasG12D mutation.

II. To identify the dose-limiting toxicities (DLT) of mesenchymal stem cell (MSC)-derived exosomes loaded with siRNA against KrasG12D (iExosomes) in metastatic PDAC patients with KrasG12D mutation.

SECONDARY OBJECTIVES:

I. Evaluate the pharmacokinetic profile of iExosomes. II. Assess the overall response rate of iExosomes in the chosen patient population.

III. Assess the disease control rate (partial response + stable disease) with therapy.

IV. Determine median progression-free survival (PFS) with this treatment. V. Determine the median overall survival (OS) with this treatment.

EXPLORATORY OBJECTIVES:

I. Evaluate optional tissue collection and serum-derived exosomes and circulating-free deoxyribonucleic acid (DNA) (cfDNA) for detection of DNA and ribonucleic acid (RNA) showing KrasG12D sequence; evaluate DNA and RNA showing KrasG12D sequence in optional tissue collection.

II. Evaluate the siRNA content in blood and optional tissue collection.

OUTLINE: This is a dose-escalation study.

Participants receive mesenchymal stromal cells-derived exosomes with KrasG12D siRNA intravenously (IV) over 15-20 minutes on days 1, 4, and 10. Treatment repeats every 14 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Participants who respond may continue 3 additional courses.

After completion of study treatment, participants are followed up at 30 days, then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed metastatic pancreatic ductal adenocarcinoma harboring KrasG12D mutation
* Patients must have documented progression or stable disease on one or more lines of systemic therapy. If stable disease, patient must have completed at least 4 months of chemotherapy with cytotoxic therapy
* KrasG12D mutation status will be informed from any previous routine molecular profiling (using commercial assays such as Foundation One, Caris, Oncomine or other) of tissue or blood. Additional KrasG12D mutation status may be confirmed using tissue biopsy or blood prior to enrolling into the trial
* ECOG (Eastern Cooperative Oncology Group) performance status of 0-1
* Absolute neutrophil count (ANC) more or equal to 1,500 cells/mm3
* Platelets more or equal to 100,000/ul
* Hemoglobin more than 9.0 g/dL
* Total bilirubin between 1 and 1.5 mg/dL
* AST (aspartate aminotransferase) and ALT (alanine transaminase) less than 2.5 x ULN (upper limit of normal)
* Alkaline phosphatase less than 2.5 x ULN
* Creatinine less than 1.5 gm/dL
* In patients with known Gilbert's syndrome, direct bilirubin less or equal to 1.5 x ULN will be used as organ function criteria, instead of total bilirubin
* Negative serum pregnancy test in women with childbearing potential (WOCBP) defined as not post-menopausal for 12 months or no previous surgical sterilization, within one week prior to initiation of treatment. WOCBP must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of study drug to minimize the risk of pregnancy. WOCBP must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of study drug to minimize the risk of pregnancy
* A male subject of fathering potential must use an adequate method of contraception to avoid conception throughout the study and for up to 12 weeks after the last dose of study drug to minimize the risk of pregnancy. If the partner is pregnant or breastfeeding, the subject must use a condom
* Patients must sign an informed consent and authorization indicating that they are aware of the investigational nature of this study and the known risks involved

Exclusion Criteria:

* Concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study such as unstable angina, myocardial infarction within 6 months, unstable symptomatic arrhythmia, uncontrolled diabetes, serious active or uncontrolled infection
* Pregnancy (positive pregnancy test) or lactation
* Known CNS (central nervous system) disease, except for treated brain metastasis. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (magnetic resonance imaging-MRI or computerized tomography-CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; gamma knife, linear accelerator [LINAC], or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to day 1 will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose Determined by Dose Limiting Toxicity | First 4 weeks of treatment
  Dose limiting toxicity graded according to the NCI CTCAE, Version 4.0
Minimal residual disease rate in high-risk patients | Up to 1 year
  Will be modeled using logistic regression.
Overall survival (OS) | Up to 1 year
  Estimated using the Kaplan-Meier product limit estimator.
Progression-free survival (PFS) | Up to 1 year
  Estimated using Kaplan-Meier product limit estimator.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Smaglo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Sall IM, Flaviu TA. Plant and mammalian-derived extracellular vesicles: a new therapeutic approach for the future. Front Bioeng Biotechnol. 2023 Sep 13;11:1215650. doi: 10.3389/fbioe.2023.1215650. eCollection 2023. PMID 37781539
- [Derived] Tang M, Chen Y, Li B, Sugimoto H, Yang S, Yang C, LeBleu VS, McAndrews KM, Kalluri R. Therapeutic targeting of STAT3 with small interference RNAs and antisense oligonucleotides embedded exosomes in liver fibrosis. FASEB J. 2021 May;35(5):e21557. doi: 10.1096/fj.202002777RR. PMID 33855751
- See also: M D Anderson Cancer Center — http://www.mdanderson.org